CLINICAL TRIAL: NCT00029757
Title: Buccal Estrogen in Toothpaste Study: Systemic Absorption of Estradiol When Administered Mixed With Toothpaste in Postmenopausal or Surgically Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR02558-1056
Record Dates: First submitted 2002-01-22; First posted 2002-01-23 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2003-12

CONDITIONS: Menopause; Postmenopause
Keywords: Surgical menopause
MeSH Terms: interventions — Estrogens

INTERVENTIONS:
Drug: Estrogen

SUMMARY:
Background: The use of estrogen in postmenopausal (or surgically menopausal) women is a common practice. Compliance is problematic in that estimates show only 1/3 of women use hormone replacement therapy (HRT) and only 30% are compliant. Estrogen has many documented benefits including symptomatic relief of hot flashes, improvement of the dry vagina and dyspareunia. Estrogen has been found to improve bone mineral density and increase the high- density lipoprotein portion of a cholesterol panel. To improve compliance and to provide an alternate method of delivery, we propose the use of estrogen which is admixed in toothpaste and propose to study the absorption, rate of build-up and rate of decline.

Hypothesis: Estrogen can potentially be absorbed systemically when toothpaste is admixed with estradiol and is applied in a timed, consistent fashion to postmenopausal or surgically postmenopausal women, not on HRT. Absorption takes place across the buccal mucosa.

Specific Aims:1) To estimate the systemic absorption of estrogen from daily use of estrogen containing toothpaste.

2) To estimate the rate of build-up of serum estrogen levels based upon daily use of toothpaste containing estrogen for eight days.

3) To estimate the rate of decline in serum estrogen levels when the use of estrogen containing toothpaste is discontinued for a week.

DETAILED DESCRIPTION:
Methods: Fifteen women ages 35-75 who are menopausal or surgically menopausal will be identified, with exclusion based on estrogen contraindications. Subjects will have blood samples taken before, during and after an eight-day course of once-daily toothpaste that is admixed with 0.5 mg estradiol. Toothpaste shall meet strict quality control standards and instructions for uniform tooth brushing shall be provided. Serum estradiol will be determined from the samples obtained. Statistical analysis shall address absorption by comparing baseline estradiol measurements with those a few hours after use. The rate of build-up will be assessed by comparing the post-use levels of estradiol at the start of a week and at the end of the week. After a week off the estrogen, the rate of decline in serum estradiol will be calculated.

ELIGIBILITY:
Postmenopausal women or surgically menopausal women, not on hormone replacement therapy for at least 3 weeks

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas--Houston Medical School, Houston, Texas, United States